CLINICAL TRIAL: NCT06431126
Title: Nature and Animal-assisted Activities for Young Adults With Autism and Social Withdrawal
Brief Title: Nature and Animal-assisted Activities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kronoberg County Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RK-997623
Record Dates: First submitted 2024-05-14; First posted 2024-05-28 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Neuropsychiatric Syndrome; Autism Spectrum Disorder
Keywords: complementary therapies; feasability; young adults
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nature and animal-assisted activities for young adults with autism (Experimental)
  Interventions: Other: Nature and animal-assisted activities

INTERVENTIONS:
Other: Nature and animal-assisted activities — Supervised activities on a farm, 2 half day/week for 12 weeks

SUMMARY:
Neuropsychiatric impairments in young adults are common and can involve social withdrawal, and difficulties in receiving support from healthcare and municipal social care services. Collaboration is needed, but knowledge gaps exist concerning effective interventions. Participation in meaningful activities, as a complement to other treatment strategies can be a step towards studies/work. The aim of the trial is to explore the feasibility of a structured nature and animal-based activity on a farm for young adults with neuropsychiatric impairments.

The intervention involves participation in nature and animal-assisted group activities, twice a week for 12 weeks. Data consists of interviews with participants prior to and after the intervention, as well as one year later. The one-year follow-up focus is on life situation, changes in everyday life and experiences of the intervention. In addition, interview-based experiences of the ordinary staff and supervisors on the farm are included. Analysis will be carried out with qualitative content analysis, as well as health-economic calculations.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years
* Autism Spectrum Disorder
* No occupation/employment/education over the last year
* Social insurance benefits
* Interest in being with animals

Exclusion Criteria:

* Ongoing active drug abuse
* Severe psychiatric comorbidity

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Attendance | 12 weeks
  Number of sessions with participation

SECONDARY OUTCOMES:
Experiences of participation | 12 weeks
  Interviews
Occupational level | 1 year
  Interview

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta Gunnarsson, PhD, Principal Investigator — Kronoberg County Council
Locations (1):
- Kronoberg County Council, Vaxjo, Sweden